CLINICAL TRIAL: NCT05659589
Title: Prognostic Role of the Uremic Toxin Indoxyl Sulfate on Vascular and Cardiac Functions During Acute Kidney Injury
Acronym: VASC-AKI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: PI2021_843_0143
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Acute Kidney Injury; Uremic; Toxemia; Vascular Dysfunction; Cardiac Dysfunction; Cardiovascular Prognosis
Keywords: Acute Kidney Injury; Uremic; Toxemia; vascular dysfunction; cardiac dysfunction; cardiovascular prognosis
MeSH Terms: conditions — Acute Kidney Injury; Toxemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: blood sample — Blood sample withdrawal will be done and serum creatinine, IS, PCS, FGF-23, Angiopoietin-2, VCAM-1, E-Selectin and Troponin will be measured.

SUMMARY:
Acute kidney injury (AKI) is a frequent disease in conventional hospital departments and in intensive care units. It's associated with a high risk to develop chronic kidney disease (CKD), even after a single small AKI episode. It's also associated with an important morbi-mortality, particularly cardiovascular (CV). Some studies have already showed a link between AKI and CV risk but pathologic mechanisms implicated are still unknown. In AKI and CKD, numerous substances, called uremic toxins (UT) are accumulating in blood. In CKD, those toxins, and particularly Indoxyl sulfate (IS), are known to have cardiac and vascular deleterious consequences. However, in AKI, whether acute accumulation of UT may trigger CV complications is unknown.

The purpose of this study is that during AKI, a high UT concentration, in particular IS, would be associated with early vascular and cardiac dysfunctions that can be characterized by the persistence of an accelerated pulse wave velocity (PWV). The main objective is to evaluate the correlation between UT concentrations (especially IS) and arterial stiffness (PWV measurement) at three months of an AKI episode in conventional hospital departments and in the intensive care unit of nephrology.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old.
* Patients hospitalized in conventional hospital departments and in intensive care units of nephrology.
* Patients with moderate to severe AKI (KDIGO 2 or 3) without dialysis.
* AKI from functional or organic aetiology

Exclusion Criteria:

* Patients with severe CKD (GFR<45ml/min/1.73 m2) or with kidney transplants.
* Patients with AKI from septic or obstructive aetiology.
* Patients with AKI from toxic aetiology whose toxic would be also responsable of cardia toxicity.
* Patients with sepsis or blood inflammation.
* Patients with severe chronic cardia dysfunction.
* Patients with arrhythmia or complete heart block.
* Patients with peripheral artery occlusive disease.
* Pregnancy.
* Patients on palliative care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change of pulse wave velocity (PWV) measurement from baseline | at 3 months

SECONDARY OUTCOMES:
Correlation between Para-cresyl Sulfate (PCS) concentration and PWV | 3 months
Correlation between Fibroblast Growth Factor 23 (FGF23) concentration and PWV | 3 months
Correlation between Fibroblast Growth Factor 23 (FGF23) concentration and arterial pressure measurement | 3 months
Correlation between Fibroblast Growth Factor 23 (FGF23) concentration and cardiac diastolic function | 3 months
Correlation between IS concentration and arterial pressure measurement | 3 months
Correlation between IS concentration and cardiac diastolic function | 3 months
Correlation between Para-cresyl Sulfate (PCS) concentration and arterial pressure measurement | 3 months
Correlation between Para-cresyl Sulfate (PCS) concentration and cardiac diastolic function | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Amiens hospital, Amiens, France

IPD SHARING:
Plan to Share IPD: No